CLINICAL TRIAL: NCT00321906
Title: Comparison of a Tacrolimus/Sirolimus/Prednisone Regimen Versus Tacrolimus/Azathioprine/Prednisone Immunosuppressive Regimen in Lung Transplantation
Brief Title: Comparison of Sirolimus and Azathioprine in Lung Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Astellas Pharma Inc (Industry); Loyola University (Other); University of Florida (Other); University of Pennsylvania (Other); Baylor College of Medicine (Other); Ochsner Health System (Other); Columbia University (Other); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14467B
Record Dates: First submitted 2006-05-02; First posted 2006-05-04 (Estimated); Results first posted 2014-02-04 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Delayed Graft Function; Acute Graft Rejection
Keywords: Rejection in lung transplant
MeSH Terms: conditions — Delayed Graft Function | interventions — Azathioprine; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azathioprine (Active Comparator): (tacrolimus,azathioprine/prednisone)
  Interventions: Drug: azathioprine
- Sirolimus (Active Comparator): tacrolimus/sirolimus/prednisone
  Interventions: Drug: sirolimus

INTERVENTIONS:
Drug: azathioprine — azathioprine 2mg/kg
  Arms: Azathioprine
Drug: sirolimus — sirolimus 2-4mg daily
  Arms: Sirolimus

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of two different anti-rejection drug regimens.

DETAILED DESCRIPTION:
This multicenter prospective, randomized controlled clinical trial compared the open label use of sirolimus with that of azathioprine in a tacrolimus-based immunosuppression regimen. Eligible patients were identified during a 90-day screening period immediately after transplantation and randomized via a computer-generated scheme. Patient randomization was stratified according to center and rejection status in the first 90 days after transplantation. All patients received IL-2 receptor antagonist induction therapy, tacrolimus, azathioprine, and corticosteroids until 90 days after transplantation. At 90 days after transplantation, patients were randomized at a 1:1 ratio to either continue azathioprine or change from azathioprine to sirolimus.

The dosing and levels of immunosuppressive medications were standardized for all patients included in this study. Tacrolimus was dosed at 0.04 mg/kg twice daily with target trough levels between 5 and 15 ng/ml, azathioprine was administered at 2 mg/kg daily with dose adjustments for leukopenia, sirolimus was initially dosed at 2 mg/day with target trough levels between 5 and 15 ng/ml, and prednisone was tapered to not more than 10 mg/day by 3 months after transplantation. All patients received induction therapy with either daclizumab or basiliximab as per the product package insert.

In addition, prophylactic antimicrobials were standardized among the participating sites. All patients with either donor and/or recipient cytomegalovirus (CMV)-positive serostatus received either intravenous ganciclovir or oral valganciclovir for a total of 90 days. Lung transplant recipients who were negative for both donor and recipient CMV serostatus received valacyclovir for 90 days. Antifungal prophylaxis was determined by each site. Pneumocystis jiroveci prophylaxis was continued throughout the study. Lipid-lowering medications were recommended according to the National Cholesterol Education Program guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Lung transplant recipients between the age of 18 and 65 years of age.
* Females who are capable of becoming pregnant must have a negative pregnancy test prior to consent. (Females of childbearing potential must be using a medically acceptable method of birth control for the duration of the study.)
* All patients must be able to give written informed consent.

Exclusion Criteria:

* White blood cell count (WBC) < 4.0/mm3
* Platelet count < 100,000/mm3
* Severe hypercholesterolemia (> 350 mg/dl) or hypertriglyceridemia (> 500 mg/dl)
* Uncontrolled systemic infection at the time of consent.
* Previous organ transplant
* Treatment with a drug within the last 30 days that has not received regulatory approval at the time of study entry or for the duration of the study (3 years).
* Use of maintenance immunosuppression other than daclizumab, tacrolimus, azathioprine, or prednisone prior to randomization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2002-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Garrity, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Result] Bhorade S, Ahya VN, Baz MA, Valentine VG, Arcasoy SM, Love RB, Seethamraju H, Alex CG, Bag R, Deoliveira NC, Husain A, Vigneswaran WT, Charbeneau J, Krishnan JA, Durazo-Arvizu R, Norwick L, Garrity E. Comparison of sirolimus with azathioprine in a tacrolimus-based immunosuppressive regimen in lung transplantation. Am J Respir Crit Care Med. 2011 Feb 1;183(3):379-87. doi: 10.1164/rccm.201005-0775OC. Epub 2010 Sep 10. PMID 20833822
- [Derived] Bhorade SM, Husain AN, Liao C, Li LC, Ahya VN, Baz MA, Valentine VG, Love RB, Seethamraju H, Alex CG, Bag R, DeOliveira NC, Vigneswaran WT, Garrity ER, Arcasoy SM. Interobserver variability in grading transbronchial lung biopsy specimens after lung transplantation. Chest. 2013 Jun;143(6):1717-1724. doi: 10.1378/chest.12-2107. PMID 23370547

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Azathioprine | Sirolimus
Started | 94 | 87
Completed | 48 | 31
Not Completed | 46 | 56
Not completed — Adverse Event | 36 | 44
Not completed — Death | 9 | 6
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azathioprine | Sirolimus | Total
Number analyzed (Participants) | 94 | 87 | 181
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [52 to 62] | 57 [48 to 60] | 57 [50 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 34 | 74
  Male | 54 | 53 | 107

OUTCOME MEASURES:

1. Primary Outcome: Acute Rejection Rate at 12 Months
Description: Raw proportion of patients that experienced acute rejection at or before 12 months.
Time Frame: 12mos
Measure: Number; unit: percentage of participants
Arm/Group | Azathioprine | Sirolimus
Number analyzed (Participants) | 94 | 87
percentage of participants | 48 | 39

2. Secondary Outcome: Acute Rejection-free Survival at 12 Months
Description: Kaplan-Meier estimate of proportion of patients that had not experienced acute rejection by 12 months. Acute rejection is defined as rejection at any of the following grades.
  Grade A0 - None With/Without Grade A1 - Minimal Grade A2 - Mild Grade A3 - Moderate
Time Frame: 12 mos
Population: The analysis population included patients who underwent at least one transbronchial biopsy.
Measure: Number; unit: percentage of participants
Arm/Group | Azathioprine | Sirolimus
Number analyzed (Participants) | 89 | 76
percentage of participants | 56 | 58

3. Secondary Outcome: Severity of Acute Rejection at 12 Months
Description: Raw proportion of patients that experienced rejection at or above grade A2 by 12 months.
  Grade A0 - None With/Without Grade A1 - Minimal Grade A2 - Mild Grade A3 - Moderate
Time Frame: 12 mos
Measure: Number; unit: percentage of participants
Arm/Group | Azathioprine | Sirolimus
Number analyzed (Participants) | 94 | 87
percentage of participants | 24 | 18

4. Secondary Outcome: Bronchiolitis Obliterans Syndrome (BOS) at 24 Months
Description: Kaplan-Meier estimate of proportion of patients that had not experienced BOS by 24 months.
Time Frame: 24 mos
Measure: Number; unit: percentage of participants
Arm/Group | Azathioprine | Sirolimus
Number analyzed (Participants) | 94 | 87
percentage of participants | 81 | 78

5. Secondary Outcome: Bronchiolitis Obliterans Syndrome (BOS) at 36 Months
Description: Kaplan-Meier estimate of proportion of patients that had not experienced BOS by 36 months.
Time Frame: 36 mos
Measure: Number; unit: percentage of participants
Arm/Group | Azathioprine | Sirolimus
Number analyzed (Participants) | 94 | 87
percentage of participants | 76 | 72

6. Secondary Outcome: Overall Survival at 12 Months
Description: Kaplan-Meier estimate of proportion of patients that survived to (i.e., had not died by) 12 months.
Time Frame: 12 mos
Measure: Number; unit: percentage of participants
Arm/Group | Azathioprine | Sirolimus
Number analyzed (Participants) | 94 | 87
percentage of participants | 97 | 97

7. Secondary Outcome: Overall Survival at 24 Months
Description: Kaplan-Meier estimate of proportion of patients that survived to (i.e., had not died by) 24 months.
Time Frame: 24 mos
Measure: Number; unit: percentage of participants
Arm/Group | Azathioprine | Sirolimus
Number analyzed (Participants) | 94 | 87
percentage of participants | 89 | 94

8. Secondary Outcome: Overall Survival at 36 Months
Description: Kaplan-Meier estimate of proportion of patients that survived to (i.e., had not died by) 36 months.
Time Frame: 36 mos
Measure: Number; unit: percentage of participants
Arm/Group | Azathioprine | Sirolimus
Number analyzed (Participants) | 94 | 87
percentage of participants | 84 | 87

ADVERSE EVENTS:
Time Frame: 3 years post-transplant
Arm/Group | Azathioprine | Sirolimus
Serious Adverse Events (participants affected / at risk) | 32/94 | 47/87
Other Adverse Events (participants affected / at risk) | 94/94 | 87/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azathioprine (N=94) | Sirolimus (N=87)
Renal insufficiency or increased creatinine level (Investigations) | 12 | 20
Anemia/Leukopenia (Blood and lymphatic system disorders) | 7 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2
Declining pulmonary function (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 6
Bacterial infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Eyelash infection (Infections and infestations) | 15 | 3
Love (Cardiac disorders) | 3 | 4
Fear of handshakes (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azathioprine (N=94) | Sirolimus (N=87)
Dyslipidemia (Metabolism and nutrition disorders) | 40 | 59
Severe hypertriglyceridemia (.500 mg/dl) (Metabolism and nutrition disorders) | 3 | 13
Abdominal pain (Gastrointestinal disorders) | 12 | 14
Nausea (Gastrointestinal disorders) | 3 | 8
Diarrhea (Gastrointestinal disorders) | 5 | 11
Renal insufficiency or increased creatinine level (Renal and urinary disorders) | 21 | 14
Diabetes Mellitus (Metabolism and nutrition disorders) | 46 | 53
Anemia/Leukopenia (Blood and lymphatic system disorders) | 26 | 19
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 15
Declining pulmonary function (Respiratory, thoracic and mediastinal disorders) | 10 | 9
Persistent acute rejection (General disorders) | 9 | 4
Thromboembolic disease (Vascular disorders) | 3 | 15
Bronchial stenosis (Respiratory, thoracic and mediastinal disorders) | 16 | 20
Pedal edema (General disorders) | 1 | 6
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Excess bleeding (Blood and lymphatic system disorders) | 1 | 5
Bacterial infection (Infections and infestations) | 31 | 38
Viral infection (Infections and infestations) | 26 | 22
Fungal infection (Infections and infestations) | 17 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes